CLINICAL TRIAL: NCT02395120
Title: Family Intervention With Caregivers of Children With Dental Needs
Brief Title: Family Access to Dentist Study
Acronym: FADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Washington (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Harvard University (Other)
Responsible Party: Principal Investigator, Suchitra Nelson, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 1-14-15; U01DE024167-01 (NIH)
Record Dates: First submitted 2015-03-17; First posted 2015-03-20 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
Keywords: Dental Care; Caregiver Illness Perception; Common Sense Model of Self-Regulation; Dental Access; Referral letter; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Standard letter (Active Comparator): Modified standard letter will be sent to caregivers.
  Interventions: Behavioral: Standard letter
- Intervention letter (Experimental): The CSM-based referral letter alone will be sent to caregivers
  Interventions: Behavioral: Intervention letter
- Reduced intervention letter (Experimental): The reduced (removing text corresponding to "timeline") CSM-based referral letter alone will be sent to caregivers.
  Interventions: Behavioral: Reduced intervention letter
- Intervention letter+DIG (Experimental): The CSM-based referral letter with the dental information guide will be sent to caregivers.
  Interventions: Behavioral: Intervention letter; Behavioral: DIG
- Reduced intervention letter+reduced DIG (Experimental): The reduced CSM-based referral letter with the reduced dental information guide will be sent to caregivers.
  Interventions: Behavioral: Reduced intervention letter; Behavioral: Reduced DIG

INTERVENTIONS:
Behavioral: Standard letter — Standard referral letter according to Ohio Department of Health Bureau guidelines. This letter is consistent with others used across the country.
  Arms: Standard letter
Behavioral: Intervention letter — Referral letter based on the Common Sense Model of Self-Regulation (CSM). The letter includes the cognitive dimensions of the CSM (identity, cause, timeline, consequences and control).
  Arms: Intervention letter; Intervention letter+DIG
Behavioral: Reduced intervention letter — Reduced (removing text corresponding to "timeline") CSM theory-based referral letter. The letter includes the remaining cognitive dimensions of the CSM (identity, cause, consequences and control).
  Arms: Reduced intervention letter; Reduced intervention letter+reduced DIG
Behavioral: DIG — Dental information guide (DIG) to reinforce/change illness perception, knowledge about dental caries, and resources to seek care. DIG is a brochure with illustrations which provides myths and facts about dental caries, hints for getting dental care, making appointments and Medicaid access, transportation and dentist availability resources.
  Arms: Intervention letter+DIG
Behavioral: Reduced DIG — Text and illustrations related to the "timeline" construct of the CSM have been removed in the reduced dental information guide.
  Arms: Reduced intervention letter+reduced DIG

SUMMARY:
The study is a multi-site, double blind, parallel arm, community-based randomized controlled trial (phase III RCT) to evaluate the effectiveness of new referral approaches to increase receipt of dental care among inner-city urban and rural elementary school children who were screened at school and have restorative treatment needs. The study has 5 arms: The experimental intervention is the use of a theoretically driven CSM referral letter alone, the letter plus a Dental Information Guide, a reduced CSM referral letter alone, or a reduced CSM referral letter plus a reduced Dental Information Guide. The control strategy is the use of a standard referral letter. All participating K-4 grade children will receive a screening at the beginning of the school year and at the study end point 7 months later to determine if the child received dental care. Due to lower than expected enrollment in both the Ohio and Washington sites, a second year of recruitment was added to include Bedford School District and East Cleveland School District (only KG and other grades if they did not enroll in the first year). The same study procedures, schedule and design was utilized for the second year of recruitment.

The primary aim is to evaluate the effectiveness of experimental (new) versus standard referral approach given to parents/caregivers in increasing receipt of dental care among their children in grades K-4. The secondary aim is to assess changes in parent/caregiver illness representation/perception and behavioral intention between enrollment (beginning of school year) and follow-up (end of school year) to understand the underlying mechanisms of the new vs. standard referral approach that result in receipt of dental care.

The hypothesis is that CSM-based interventions will increase receipt of dental care compared to the standard referral letter.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate the effectiveness of new referral approaches to increase receipt of dental care among inner-city urban and rural elementary school children who were screened at school and have restorative treatment needs. The primary outcome is the assessment of dental care receipt through dental exams. The secondary outcomes are change in caregiver illness perception, measured through the IPQ-RD, and behavioral intention measured through items in the caregiver questionnaire.

Study Design:

The study will utilize a multi-site, double-blind, parallel arm, community-based randomized trial design. The experimental intervention will be based upon the Common Sense Model of Self-Regulation (CSM) to address parent/caregiver illness perception and navigation of resources to increase receipt of dental care during a 7-month follow-up period for children with restorative dental needs. In this five arm study the new CSM theory-driven referral letter alone, the new CSM referral letter and Dental Information Guide (DIG), the new CSM theory-driven reduced referral letter alone, and the new CSM theory-driven reduced referral letter and reduced Dental Information Guide (DIG) will each be compared to a standard referral letter to increase receipt of dental care among inner-city urban African American, and rural Hispanic and White elementary school children.

Participants:

Subjects will be parents/caregivers and their children in grades K-4 in one of four school districts; East Cleveland City School District (OH), Cowlitz County School Districts (WA), Lewis County School Districts (WA), and Bedford (OH). The study will be offered to all caregivers and their children including those children with special health care needs. At the Ohio site, only English-speaking caregivers and their children will be enrolled while both English- and Spanish-speaking caregivers and their children will be included at the Washington site. At the beginning of the school year dental screening, primary caregivers will be randomized if their child has a tooth with an International Caries Detection and Assessment System (ICDAS) active lesion score of 2 or greater. Caregivers with multiple children in K-4 will receive the same intervention assignment. The second year of recruitment included Bedford School District in Ohio and East Cleveland School District KG and other grade families if they did not enroll in the first year.

Procedures:

Caregivers will be recruited at the beginning of the school year and complete baseline forms (consent form, Illness Perception Questionnaire-Revised for Dental (IPQ-RD) questionnaire, and caregiver questionnaire) prior to dental screening and randomization. Children in K-4 whose parents have consented will receive a screening exam in early October 2015 (October 2016 for the second year of recruitment). After screening exams, eligible caregivers of children with restorative referrals will be randomized into one of five study arms. Different referral letter with/without Dental Information Guide according to study arms will be sent home with the child on the day of screening and mailed to the caregiver address within 24 hours.

Caregivers will be followed at 2 time points: 2 weeks after the receipt of the intervention letter and 2 weeks prior to the final (exit) study visit examinations in May 2016 (May 2017 for the second year of recruitment)-approximately 7 months after the initial dental exam. At both time points caregivers will complete the IPQ-RD and the caregiver questionnaire. A small sub-sample of 60 caregivers will be randomly sampled from three arms (standard letter, intervention letter, and intervention letter+DIG) to complete the IPQ-RD 1 month after enrollment for fidelity purposes. All questionnaires will be mailed to the home address and asked to be returned to the class-room teacher or the outreach staff. Further, outreach staff will ensure that the caregivers received and returned the materials through follow-up calls. Children will have a follow-up dental exam in May 2016 (May 2017 for the second year of recruitment).

Analysis Plan:

Primary Statistical Analysis: Descriptive statistics will include frequencies (categorical variables) and means (continuous variables) of baseline covariates among the five intervention groups. Chi-square tests (for categorical variables) and t-tests (for continuous variables) will be performed to test for group differences (by site and overall). In our primary analysis, we will fit multivariate generalized linear (specifically, logistic regression) models with dental care receipt as the (binary) outcome and the child as the unit of analysis (as receipt of dental care will be determined for each child). A generalized estimating equations (GEE) approach (with an exchangeable working correlation structure) will be used to allow for correlations among multiple children for a given caregiver. Secondarily, we will fit a model with a site by intervention group interaction, and the latter will be tested to formally assess possible intervention effect heterogeneity over sites.

We will also consider working correlation structures (e.g., alternating logistic regressions) that allow for second-level clusters, namely schools (within which the first-level cluster, caregiver, is nested). We will determine final models based on the quasi-likelihood information criterion (QIC). Intervention (and other covariate) effects will be tested using generalized score statistics.

Analysis of Secondary Outcomes (Questionnaire data): Summary statistics (including means and standard errors) for questionnaire responses for both the IPQ-RD and behavioral intention items within the caregiver questionnaire will be calculated by site and intervention group. This will be done for the overall questionnaire (IPQ-RD and behavioral intention), for each of the five IPQ-RD cognitive constructs, and the two behavioral intention questions. Analyses will be done by site and overall (controlling for site). A summary measure approach, based on the mean questionnaire response, will be used to compare questionnaire outcomes across intervention groups, for the overall questionnaire and by construct. Specifically, for each construct (or overall) a linear regression model will be used with the mean response as the dependent variable, and intervention group indicators and selected baseline (control) covariates as independent variables. Inferences (that is, p-values and confidence intervals) will be performed assuming summary measures are normally distributed. This assumption will be tested using the Shapiro-Wilk statistic and if violated a suitable transformation of the summary measure used or a nonparametric approach (e.g., using ranks of the summary measures) conducted.

Missing Data:

In the event of missing questionnaire responses, we will first assess whether the data are missing completely at random (MCAR), that is, whether missingness for a given item is dependent only on participant baseline characteristics and not further on any other item responses. This will be done using a generalized estimating equations (GEE) approach, that is, by fitting a multivariate generalized linear (e.g., logistic regression) model to missing data indicators for each item, including as explanatory variables selected baseline covariates and other item responses, and testing for an effect of the latter.

If the MCAR assumption is deemed reasonable (no significant effect found), we will conduct the above regression analyses with mean outcomes based on available data. A weighted analysis (that is, regression with the use of the weighted least squares criterion) will be conducted to adjust for differential missingness (thus, non-homogeneous summary measure variances) among participants. If the MCAR assumption is found to be violated we will use a multiple imputation approach (in conjunction with the summary measure approach) using a suitable imputation model (i.e., using other item responses). For each construct (or overall) we will perform an F-test for a difference in the mean summary measure among the three intervention groups, and obtain nominal 95% confidence intervals for pairwise mean differences. If necessary, we will include a random effect for school.

Data Management:

Data for this study are captured using examinations, forms, questionnaires, and audio recordings. Study data will be collected and stored using the REDCap platform. REDCap is a secure, web-based application designed to support remote data capture for research studies, providing: 1) an intuitive interface for validated data entry, 2) audit trails for tracking data manipulation and export procedures, 3) automated export procedures for seamless data downloads to common statistical packages, and 4) procedures for importing data from external sources.

Study forms will be completed by study personnel on paper, and subsequently entered into REDCap by study staff. Because randomization is contingent upon the computer, no paper randomization forms will be completed. Paper forms will be securely stored in a locked file cabinet at both sites when they are not in use. Completed paper forms will be transferred between sites via courier or other secure document service. Similarly, questionnaires used in the study (IPQ-RD, Caregiver Questionnaire) will be completed by subjects on paper sheets and returned to Outreach Workers in each school. Study staff will enter the information into the database. All data forms, questionnaires will be entered into database stored in a secure password protected computer. Recorded audios will be stored in secured/locked cabinets in one of the Project Coordinators' offices.

Dental examination and study questionnaire data will be reviewed for accuracy and completeness after each study visit. The Outreach Workers will review the questionnaires after the participants have completed them, and the Project Coordinators and the Data and Statistics Team will do a final review after the documents have been transmitted. An annual report (or as requested by the DSMB or NIDCR Program Official) will also be generated for sharing progress of the study.

The Data & Statistics Team will generate regular reports showing enrollment and potential data anomalies, which will be sent to PIs, Project Coordinators, and other relevant study staff. The Data Manager will work with the PIs at each site to resolve any data anomalies that arise during recruitment. The Data & Statistics Team will also respond to data queries generated by the PIs, Project Coordinators, or other study staff.

Statistical analyses and summary reports will be generated by the study Biostatistician during the course of the study. At the end of the study, the study Biostatistician will conduct analyses of the data and assist in preparation of study publications and presentations. The Data Manager will provide technical and data support for the Biostatistician throughout the study.

ELIGIBILITY:
Inclusion Criteria: (parents/caregivers and their children)

* Provide signed and dated consent form (also assent form for children 7 and older)
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female child, grades K-4
* Child in good general health as evidenced by parent report (including children with special health care needs)
* Based on the beginning of the school year dental screening, caregivers will be randomized if their child has tooth with an International Caries Detection and Assessment System (ICDAS) active lesion score of ≥ 2

Exclusion Criteria: (parents/caregivers)

* Illiterate
* Non-English speaking (in East Cleveland Public Schools)
* Under 18 years of age

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1305 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Nelson, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelson S, Milgrom P, Albert JM, Selvaraj D, Cunha-Cruz J, Curtan S, Copeland T, Heima M, Rothen M, Beck G, Ferretti G, Riedy C. Randomized Trial Based on the Common-Sense Model of Self-regulation to Increase Child Dental Visits. JDR Clin Trans Res. 2019 Oct;4(4):323-332. doi: 10.1177/2380084419830662. Epub 2019 Feb 22. PMID 30931720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children in grades K-4 and their caregivers were recruited from six school districts in Ohio and Washington (14 schools) in school years 2015/2016 and 2016/2017 to participate in the baseline dental screening at the beginning of the year (phase 1). Those with untreated cavities were eligible to participate in the clinical trial phase of the study (phase 2).
Pre-assignment Details: Out of 1,584 children screened, 694 had untreated cavities that needed restorative care. Caregivers were randomized if their child had any tooth with an International Caries Detection and Assessment System (ICDAS) active lesion score ≥2. The caregivers (n=611) and their children (694) were randomized to the 5 arms of the study. 97children transferred or were absent for the baseline dental exam days.
Period: Overall Study
Arm/Group | Intervention Letter | Intervention Letter+DIG | Reduced Intervention Letter | Reduced Intervention Letter+Reduced DIG | Standard Letter
Started (Caregivers and Children) | 400 (Caregivers and Children) | 398 (Caregivers and Children) | 43 (Caregivers and Children) | 63 (Caregivers and Children) | 401 (Caregivers and Children)
Started-Caregivers (Caregivers (primary caregiver of family)) | 188 | 188 | 20 | 28 | 187
Started-Children (Children (can be multiple children of caregiver)) | 212 | 210 | 23 | 35 | 214
Completed-Caregivers (Caregivers (primary caregiver of family)) | 161 | 159 | 17 | 25 | 164
Completed-Children (Children (can be multiple children of caregiver)) | 182 | 177 | 20 | 32 | 186
Completed (Caregivers and Children) | 343 (Caregivers and Children) | 336 (Caregivers and Children) | 37 (Caregivers and Children) | 57 (Caregivers and Children) | 350 (Caregivers and Children)
Not Completed | 57 | 62 | 6 | 6 | 51
Not completed — Missed follow-up dental exam | 57 | 62 | 6 | 6 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Letter | Intervention Letter+DIG | Reduced Intervention Letter | Reduced Intervention Letter+Reduced DIG | Standard Letter | Total
Number analyzed (Participants) | 400 | 398 | 43 | 63 | 401 | 1305
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The analysis population differs from the overall population due to missing data and including only the age of the caregivers. The age of the children was not collected as inclusion criteria was based on the grade of the child (K-4), not on age.
  years
    Caregiver Age: number analyzed (Participants) | 161 | 159 | 17 | 25 | 164 | 526
    Caregiver Age | 34.06 (7.09) | 34.63 (9.78) | 31.46 (3.5) | 34.22 (8.16) | 32.55 (8.15) | 33.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population differs from the overall population due to missing data for some participants.
  Participants
    Caregiver Sex: number analyzed (Participants) | 179 | 180 | 17 | 23 | 179 | 578
    Caregiver Sex: Female | 165 | 166 | 16 | 21 | 166 | 534
    Caregiver Sex: Male | 14 | 14 | 1 | 2 | 13 | 44
    Children Sex: number analyzed (Participants) | 196 | 202 | 20 | 26 | 202 | 646
    Children Sex: Female | 110 | 121 | 11 | 12 | 107 | 361
    Children Sex: Male | 86 | 81 | 9 | 14 | 95 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population is reported separately for caregivers and children.
  Participants
    Caregiver Ethnicity: number analyzed (Participants) | 188 | 188 | 20 | 28 | 187 | 611
    Caregiver Ethnicity: Hispanic or Latino | 21 | 16 | 2 | 2 | 11 | 52
    Caregiver Ethnicity: Not Hispanic or Latino | 79 | 83 | 8 | 12 | 85 | 267
    Caregiver Ethnicity: Unknown or Not Reported | 88 | 89 | 10 | 14 | 91 | 292
    Children Ethnicity: number analyzed (Participants) | 212 | 210 | 23 | 35 | 214 | 694
    Children Ethnicity: Hispanic or Latino | 23 | 19 | 4 | 4 | 25 | 75
    Children Ethnicity: Not Hispanic or Latino | 89 | 89 | 8 | 15 | 88 | 289
    Children Ethnicity: Unknown or Not Reported | 100 | 102 | 11 | 16 | 101 | 330
Race (NIH/OMB) [Count of Participants; unit: Participants] — Caregivers Population: The analysis population is reported separately for caregivers and children.
  Participants
    Caregiver Race: number analyzed (Participants) | 188 | 188 | 20 | 28 | 187 | 611
    Caregiver Race: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
    Caregiver Race: Asian | 1 | 1 | 0 | 0 | 0 | 2
    Caregiver Race: Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2 | 4
    Caregiver Race: Black or African American | 90 | 88 | 9 | 11 | 92 | 290
    Caregiver Race: White | 47 | 54 | 6 | 7 | 56 | 170
    Caregiver Race: More than one race | 5 | 8 | 1 | 2 | 7 | 23
    Caregiver Race: Unknown or Not Reported | 44 | 35 | 4 | 8 | 30 | 121
    Children Race: number analyzed (Participants) | 202 | 200 | 20 | 26 | 198 | 646
    Children Race: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
    Children Race: Asian | 1 | 1 | 0 | 0 | 0 | 2
    Children Race: Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2 | 4
    Children Race: Black or African American | 97 | 90 | 11 | 13 | 82 | 293
    Children Race: White | 51 | 50 | 5 | 8 | 48 | 162
    Children Race: More than one race | 5 | 11 | 2 | 0 | 8 | 26
    Children Race: Unknown or Not Reported | 47 | 46 | 2 | 5 | 58 | 158
Education [Count of Participants; unit: Participants] — Population: Data is provided for caregivers. Children were all in grades K-4. The analysis population differs from the overall population due to missing data for some participants.
  Participants
    Greater than high school: number analyzed (Participants) | 155 | 166 | 15 | 16 | 161 | 513
    Greater than high school | 82 | 89 | 8 | 9 | 75 | 263
    Less than or equal to high school: number analyzed (Participants) | 155 | 166 | 15 | 16 | 161 | 513
    Less than or equal to high school | 73 | 77 | 7 | 7 | 86 | 250
Marital Status [Count of Participants; unit: Participants] — Population: Data is provided for caregivers. The Analysis population also differs from the overall population due to missing data for some participants.
  Participants
    Married: number analyzed (Participants) | 156 | 167 | 15 | 16 | 163 | 517
    Married | 50 | 42 | 5 | 4 | 45 | 146
    Other: number analyzed (Participants) | 156 | 167 | 15 | 16 | 163 | 517
    Other | 106 | 125 | 10 | 12 | 118 | 371

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Receipt of Dental Care-restoration or Extraction of at Least One Tooth at Final Exam
Description: The primary outcome was receipt of dental care based on a change in the child's oral health status, as determined by clinical examinations between baseline screening (beginning of schoolyear) and follow-up at study exit (end of school year). A child was classified as having received dental care if she or he had any tooth at follow-up with an ICDAS sealant code (1 or 2),restoration code (3 to 8), or extraction code (X), previously identified at baseline via an active ICDAS lesion code ≥2.
Time Frame: Between baseline and follow-up (7 months after baseline)
Population: Participants analyzed for the primary outcome are children.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Letter | Intervention Letter+DIG | Reduced Intervention Letter | Reduced Intervention Letter+Reduced DIG | Standard Letter
Number analyzed (Participants) | 182 | 177 | 20 | 32 | 186
Participants | 68 | 76 | 8 | 14 | 71
Statistical Analysis 1: Comparison: Intervention Letter vs Intervention Letter+DIG vs Reduced Intervention Letter vs Reduced Intervention Letter+Reduced DIG vs Standard Letter; Test type: Superiority; p < 0.05, Regression, Logistic — We addressed the issue of multiple testing, both multiple comparisons and multiple sites, using a gatekeeper approach. The use of 0.05 alpha level for each test maintained a 0.05 family-wise alpha level for the six tests (three at each site); Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.21 to 3.08]; The primary outcome analysis utilized generalized estimating equations (GEE) with a logit link for the binary dental care receipt outcome. The GEE analysis was conducted using dental care receipt outcomes as restorative care alone (ICDAS codes ≥3), as well as combined preventive (i.e. sealants) and restorative care (ICDAS codes ≥1). Models were fit separately to the overall data (all sites combined), the combined EC and WA sites (based on our original plan of two predominantly low-income school districts), and the BD schools alone. Each model included, as covariates, indicator variables for intervention, site (except for the model with BD alone), child grade, and caregiver demographic variables (race, education, marital status). Corresponding estimated odds ratios and 95% Confidence Intervals were computed

2. Secondary Outcome: Change in Illness Perception Assessed by IPQ-RD
Description: Change in the overall Illness Perception Questionnaire-Revised for Dental (IPQ-RD) mean score from baseline to the final data collection timepoint. The IPQ-RD is a 32 item instrument with scale responses going from 1 to 5 (strongly agree to strongly disagree) with strongly agree and agree being an accurate response. This was converted to an accurate (1,2) and inaccurate (3,4,5) dichotomous variable for each IPQ-RD item. A proportion of accurate responses was calculated for each participant (i.e. number of accurate responses divided by the total number of IPQ-RD items). The mean proportion of accurate responses was calculated as the average for the total number of participants who completed the IPQ-RD instrument. Since a lower score on the IPQ-RD is an accurate response, the difference of baseline minus final follow-up results in a negative score meaning an improved score from baseline.
Time Frame: Between baseline and final follow-up
Population: Analysis was completed for caregivers who completed the final follow-up IPQ-RD Questionnaire.
Measure: Mean (Standard Deviation); unit: mean proportion of accurate responses
Arm/Group | Intervention Letter | Intervention Letter+DIG | Reduced Intervention Letter | Reduced Intervention Letter+Reduced DIG | Standard Letter
Number analyzed (Participants) | 86 | 94 | 13 | 12 | 98
mean proportion of accurate responses | -2.65 (18.24) | -2.79 (19.09) | -1.96 (18.80) | 1.96 (25.62) | -1.10 (19.51)

3. Secondary Outcome: Number of Caregivers With Change in Behavioral Intention
Description: Behavioral intention is measured by the percent of "yes" responses to the item "I want to take my child to the dentist" and "I plan to take my child to the dentist". Caregivers who have taken the child to the dentist will skip this question at follow-up.
Time Frame: Final follow-up (7 months)
Population: Analysis was done for caregivers completing the question at the final timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Letter | Intervention Letter+DIG | Reduced Intervention Letter | Reduced Intervention Letter+Reduced DIG | Standard Letter
Number analyzed (Participants) | 33 | 38 | 2 | 6 | 40
Participants | 25 | 34 | 1 | 5 | 33

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | Intervention Letter | Intervention Letter+DIG | Reduced Intervention Letter | Reduced Intervention Letter+Reduced DIG | Standard Letter
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/398 | 0/43 | 0/63 | 0/401
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/398 | 0/43 | 0/63 | 0/401
Other Adverse Events (participants affected / at risk) | 0/400 | 0/398 | 0/43 | 0/63 | 0/401

LIMITATIONS AND CAVEATS:
We were not able to recruit the full sample size of 660 parents/caregivers for 80% power, due to lower-than-expected school enrollment.

Although examiners were trained and calibrated, it was difficult to detect tooth-colored fillings and sealants. So, our outcomes may have been underestimated in all arms.

Since our outcomes were clinically determined, it is possible that parents may have taken their child to the dentist but did not complete all necessary treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT02395120/Prot_SAP_000.pdf